CLINICAL TRIAL: NCT06005298
Title: Alcohol Misuse, Gut Microbial Dysbiosis and PrEP Care Continuum: Application and Efficacy of SBIRT Intervention (SEAL)
Brief Title: Alcohol Misuse, Gut Microbial Dysbiosis and PrEP Care Continuum: Application and Efficacy of SBIRT Intervention
Acronym: SEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirish S Barve (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Shirish S Barve, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22.0606; 1R01AA030485-01 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2023-08-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Use Disorder; Risk Behavior, Health; Dysbiosis; HIV Infections
Keywords: PrEP; Alcohol; SBIRT
MeSH Terms: conditions — Alcoholism; Health Risk Behaviors; Dysbiosis; HIV Infections | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AUDIT <8 (No Intervention): Participants whose audit score is less than eight are assigned to this arm. AUDIT is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, dependence, and experience of alcohol-related harm. AUDIT <8 is non-hazardous.
- AUDIT >8 + SBIRT (Experimental): This is an experimental arm, and AUDIT >8 is hazardous. The goal is to make connections on the impact of the SBIRT intervention on PrEP engagement and alcohol use among the participants to create a full picture of the impact of the intervention on groups exhibiting different types of alcohol use.
  Interventions: Behavioral: Screening, Brief Intervention, Referral to Treatment (SBIRT)
- AUDIT > 8 NO SBIRT (No Intervention): This is NOT an experimental arm, despite an AUDIT score > 8.

INTERVENTIONS:
Behavioral: Screening, Brief Intervention, Referral to Treatment (SBIRT) — SBIRT has been defined by SAMHSA as a comprehensive, integrated, public health approach to the delivery of early intervention for individuals with risky alcohol and drug use and the timely referral to more intensive substance abuse treatment for those who have substance abuse disorders. There is consensus that a comprehensive SBIRT model includes screening, brief intervention/brief treatment, and referral to treatment. In addition there are following characteristics:
  * It is brief (e.g., typically about 5-10 minutes for brief interventions; about 5 to 12 sessions for brief treatments)
  * The screening is universal.
  * One or more specific behaviors related to risky alcohol and drug use are targeted.
  * The services occur in a public health non-substance abuse treatment setting.
  * It is comprehensive (comprised of screening, brief intervention/treatment, and referral to treatment).
  * Strong research or experiential evidence supports the model's effectiveness.
  Arms: AUDIT >8 + SBIRT

SUMMARY:
This randomized control trial study among Pre-exposure prophylactic users (PrEP) aims to learn and determine the efficacy of Screening, brief intervention, and referral to treatment (SBRIT) in reducing the risk of alcohol use. The main questions it aims to answer are:

1. How alcohol use impacts the PrEP continuum and to understand how early intervention and treatment approach affects alcohol use and PrEP adherence.
2. Investigate the effectiveness of the SBIRT intervention in preventing hazardous alcohol use and its impact on gut dysbiosis in PrEP users.
3. To determine alterations in the gut microbiome (dysbiosis), intestinal homeostasis, systemic inflammation, and markers of liver disease associated with hazardous alcohol use among PrEP users.

DETAILED DESCRIPTION:
The study pursues a randomized control trial (RCT) with persons who use pre-exposure prophylaxis (PrEP) to determine the efficacy of SBIRT (Screening, Brief Intervention, & Referral to Treatment) in reducing the risk of alcohol drinking and associated pathogenic changes in the gut liver axis.

Participants in this study will attend visits at 3 months, 6 months,s and 12 months for about 60 to 90 minutes. These visits may include filling out a survey, participating in an interview, meeting with an SBIRT interventionist, and providing the aforementioned samples: Blood, urine, stool, saliva, oral and vaginal, if applicable.

This study will use a syndemic approach to expand the HIV/AIDS prevention toolkit among populations impacted by alcohol with a range of patterns of episodic and long-term use and associated behavioral and biological risks for HIV acquisition.

Specifically, the team will execute a randomized control trial among Pre-Exposure Prophylaxis (PrEP) users demonstrating heightened alcohol use to test the effectiveness of the Screening, Brief Intervention, & Referral to Treatment (SBIRT) intervention to reduce alcohol use and examine the subsequent impact on the gut microbiome compared to individuals receiving treatment as usual and PrEP users not demonstrating elevated alcohol use. Finally, we will employ qualitative methods (in-depth interviews) and analysis to understand decision-making factors influencing PrEP adherence and alcohol use over time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years
* Confirmation of seronegative HIV, Hep B, and Hep C status
* PrEP users
* English-speaking or Spanish speaking
* Cognitively competent to provide consent
* Attend a participating healthcare facility

Exclusion Criteria:

* Inability to consent
* Existing diagnosis of major psychiatric illness
* Unstable medical conditions (e.g., cancer)
* Taking immunosuppressants or Chemotherapy
* Taking daily antibiotics or probiotics
* Severe gastrointestinal/liver disease
* Autoimmune disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-10-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Hazardous Alcohol use | baseline, 3 months, 6 months, 12 months
  Hazardous alcohol use in the experimental group (SBIRT) will be compared to the control group (treatment as usual).
Subjects AUDIT test | baseline, 3 months, 6 months, 12 months
  This will be measured by the Alcohol Use Disorders Identification Test (AUDIT), which is an alcohol screening instrument.
Subjects TLFB review | baseline, 3 months, 6 months, 12 months
  TLFB / Timeline Followback, which involves asking participants to retrospectively estimate their alcohol use 7 days to 2 years prior to the interview date.
Subjects TAPS tool | baseline, 3 months, 6 months, 12 months
  TAPS Tool / The Tobacco, Alcohol, Prescription medications, and other Substance Tool, which is a screening and assessment tool for alcohol use in the past year.
Number of Patients with Gut Microbial alpha diversity measured by the Shannon index | baseline, 3 months, 6 months, 12 months
  Another significant primary outcomes for this aim is gut microbial alpha diversity measured by the Shannon index.
  Among all PrEP users, the comparison will be done between those who drink alcohol with those who do not drink alcohol in terms of the Shannon index. This will be analyzed using stool samples.
Number of Patients with Gut Microbial alpha diversity measured by abundance of bacteria | baseline, 3 months, 6 months, 12 months
  The primary outcome for this aim- Gut microbial alpha diversity measurement using the abundance of bacteria family Lachnospiraceae.
  This involves transforming the relative abundance (RA) of Lachnospiraceae during logit transformation to expand the RA. This will be analyzed using stool samples.
Number of Patients reaching PrEP adherence by Tenofovir Urine Test | baseline, 3 months, 6 months, 12 months
  PrEP adherence in the experimental group (SBIRT) will be compared to the control group (treatment as usual). This will be measured using a single-item measure using a Tenofovir Urine Test.

SECONDARY OUTCOMES:
Number of Patients reporting self-efficacy related to PrEP or confidence in one's ability to carry out behaviors important to PrEP adherence | baseline, 3 months, 6 months, 12 months
  Self-efficacy related to PrEP or confidence in one's ability to carry out behaviors important to PrEP adherence in the experimental group (SBIRT) will be compared to the control group (treatment as usual). This will be measured by the PrEP self-efficacy scale.
Number of Patients reporting PrEP stigma by PrEP Stigma Likert Scale | baseline, 3 months, 6 months, 12 months
  PrEP stigma in the experimental group (SBIRT) will be compared to the control group (treatment as usual).
Number of Patients reporting self-efficacy related to abstaining from alcohol by AASE / Alcohol Abstinence Self-Efficacy Scale. | baseline, 3 months, 6 months, 12 months
  Self-efficacy related to abstaining from alcohol will increase in the experimental group (SBIRT) compared to the control group (treatment as usual).
Number of Patients reporting use of other illicit drugs by the ASSIST (version 2.0) / Alcohol, Smoking and Substance Involvement Screening Test | baseline, 3 months, 6 months, 12 months
  Use of other illicit drugs will decrease in the experimental group (SBIRT) compared to the control group (treatment as usual). This will be measured by the ASSIST (version 2.0) / Alcohol, Smoking and Substance Involvement Screening Test which is a screening instrument for Cannabis, Cocaine, Prescription Stimulants, Methamphetamine, Inhalants, Sedatives, Hallucinogens, Street Opioids, Prescription Opioids, other drugs, the TLFB / Timeline Followback, which involves asking participants to retrospectively estimate their illicit drug use 7 days to 2 years prior to the interview date, and the TAPS Tool / The Tobacco, Alcohol, Prescription medications, and other Substance Tool, which is a screening and assessment tool for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year.
Number of Patients reporting Sense of hope as evidenced by improved sense of goal directed energy and/or planning to accomplish goals m | baseline, 3 months, 6 months, 12 months
  Sense of hope will increase in the experimental group (SBIRT) compared to the control group (treatment as usual). This will be measured by the Adult Hope Scale (AHS).
Number of Patients reporting Symptoms of depression | baseline, 3 months, 6 months, 12 months
  Symptoms of depression will decrease in the experimental group (SBIRT) compared to the control group (treatment as usual). This will be measured by the CES-D / Center for Epidemiologic Studies Depression Scale.
Number of Patients reporting Symptoms of anxiety | baseline, 3 months, 6 months, 12 months
  Symptoms of anxiety will decrease in the experimental group (SBIRT) compared to the control group (treatment as usual). This will be measured by the CESA / Center for Epidemiologic Studies Anxiety Scale.
Number of Patients with Gut microbiome/bacterial composition at the genera level, and functional characteristics of genes for bacterial populations | baseline, 3 months, 6 months, 12 months
  Secondary outcomes from gut microbiome evaluation will be bacterial composition at the genera level, and functional characteristics of genes for bacterial populations. This will be analyzed using stool samples.
Number of Patients with Immune Activation, Inflammation and liver injury related outcomes | baseline, 3 months, 6 months, 12 months
  Secondary outcomes from plasma/blood samples will be i) Intestinal fatty acid binding protein (IFABP) and lipopolysaccharide (LPS) for gut permeability and microbial translocation; ii) sCD14 and inflammatory cytokines including TNFα, IL-1β, MCP-1, IL-8, IL-6 for immune activation and inflammation and iii)AST, ALT and CK18 for liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Barve, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumenthal J, Pasipanodya EC, Jain S, Sun S, Ellorin E, Morris S, Moore DJ. Comparing Self-Report Pre-Exposure Prophylaxis Adherence Questions to Pharmacologic Measures of Recent and Cumulative Pre-Exposure Prophylaxis Exposure. Front Pharmacol. 2019 Jul 5;10:721. doi: 10.3389/fphar.2019.00721. eCollection 2019. PMID 31333454
- [Result] Higgins-Biddle JC, Babor TF. A review of the Alcohol Use Disorders Identification Test (AUDIT), AUDIT-C, and USAUDIT for screening in the United States: Past issues and future directions. Am J Drug Alcohol Abuse. 2018;44(6):578-586. doi: 10.1080/00952990.2018.1456545. Epub 2018 May 3. PMID 29723083
- [Result] Conigrave KM, Hall WD, Saunders JB. The AUDIT questionnaire: choosing a cut-off score. Alcohol Use Disorder Identification Test. Addiction. 1995 Oct;90(10):1349-56. doi: 10.1046/j.1360-0443.1995.901013496.x. PMID 8616463
- [Result] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Result] Humeniuk R, Henry-Edwards S, Ali R, Poznyak V, Monteiro MGea. The Alcohol, Smoking and Substance involvement Screening Test (ASSIST): manual for use in primary care. Geneva, Swizterland World Health Organization;2010.
- [Result] Zhang W, O'Brien N, Forrest JI, Salters KA, Patterson TL, Montaner JS, Hogg RS, Lima VD. Validating a shortened depression scale (10 item CES-D) among HIV-positive people in British Columbia, Canada. PLoS One. 2012;7(7):e40793. doi: 10.1371/journal.pone.0040793. Epub 2012 Jul 19. PMID 22829885
- [Result] Ghare S, Singhal R, Bryant V, Gautam S, Tirumala CC, Srisailam PK, Reyes-Vega A, Ghooray D, McClain CJ, Hoffman K, Petrosino J, Bryant K, Govind V, Cohen R, Cook RL, Barve S. Age-Associated Gut Dysbiosis, Marked by Loss of Butyrogenic Potential, Correlates With Altered Plasma Tryptophan Metabolites in Older People Living With HIV. J Acquir Immune Defic Syndr. 2022 Feb 1;89(Suppl 1):S56-S64. doi: 10.1097/QAI.0000000000002866. PMID 35015746
- [Result] Fulcher JA, Li F, Cook RR, Zabih S, Louie A, Okochi H, Tobin NH, Gandhi M, Shoptaw S, Gorbach PM, Aldrovandi GM. Rectal Microbiome Alterations Associated With Oral Human Immunodeficiency Virus Pre-Exposure Prophylaxis. Open Forum Infect Dis. 2019 Oct 29;6(11):ofz463. doi: 10.1093/ofid/ofz463. eCollection 2019 Nov. PMID 32258202
- [Result] Dube MP, Park SY, Ross H, Love TMT, Morris SR, Lee HY. Daily HIV pre-exposure prophylaxis (PrEP) with tenofovir disoproxil fumarate-emtricitabine reduced Streptococcus and increased Erysipelotrichaceae in rectal microbiota. Sci Rep. 2018 Oct 12;8(1):15212. doi: 10.1038/s41598-018-33524-6. PMID 30315206
- [Result] Perler BK, Reinhart EM, Montgomery M, Maynard M, Shapiro JM, Belenky P, Chan PA. Evaluation of the Microbiome in Men Taking Pre-exposure Prophylaxis for HIV Prevention. AIDS Behav. 2021 Jul;25(7):2005-2013. doi: 10.1007/s10461-020-03130-7. Epub 2021 Jan 4. PMID 33394167